CLINICAL TRIAL: NCT00221806
Title: Randomised Study Comparing Endothelialised Prosthesis and Autologous Vein for Under Knee Revascularisation With Femoro Popliteal Bypass. ePTFE
Brief Title: Comparison of Two Under Knee Lower Limb Bypass Types:Endothelialised Prosthesis Versus Autologous Vein Graft
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government); W.L.Gore & Associates (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9256-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Arteritis
Keywords: Arteritis, femoro popliteal bypass, endothelialised prosthesis, saphenous vein graft, permeability, Doppler echography
MeSH Terms: conditions — Arteritis

INTERVENTIONS:
Device: endothelialised prosthesis

SUMMARY:
The aim of this project is to improve the hemocompatibility of vascular prosthesis with a complete covering of its endoluminal surface with autologous endothelial cells. The objective is to obtain a better bypass permeability with arterial prosthesis replacing low diameter vessels in lower limbs

DETAILED DESCRIPTION:
Physiological vascular endothelium is an hemocompatible and thrombus resistant surface and none of the materials used for revascularisation owns these properties. The aim of this project is to improve the hemocompatibility of vascular prosthesis with a complete covering of their endoluminal surface with autologous endothelial cells. This strategy, that plans to associate an artificial component of synthetic origin and cellular component is a bioartificial vascular substitute concept. First results obtained by an austrian team are really encouraging (with more than 100 patients during last 10 years). Thus, the main objective of this study is to compare efficacy in terms of grafts with endothelialised PTFE prosthesis with great saphenous autologous vein graft for under knee arterial popliteal revascularisation of lower limbs.

This is a phase III, randomised equivalent trial. It is open labelled, with 2 parallel well balanced groups. Forty patients will be randomised. A short segment of the cephalic vein will be cut and some blood will be sampled in patients randomised in the ePTFE group. Endothelial cells of the cephalic vein will be isolated, cultured, with autologous serum, and then amplified before sowing of the internal face of PTFE prosthesis, previously covered with a biological glue clinically validated. Before prosthesis implantation, systematic quality controls will be performed. Implantation will be planned 3 weeks after venous sampling. Eventual failure of cellular culture or prosthesis covering will lead to an autologous vein graft. People randomised in the second group will receive an autologous saphenous vein graft.

The primary outcome is to demonstrate the equivalence of time dependent permeability rate between endothelialized PTFE and autologous vein graft. Equivalence between both technics would allow to preserve autologous saphenous vein for later distal bypasses (where it is the best technic) or for coronary bypasses.

ELIGIBILITY:
Inclusion Criteria:

Age above 18, male or female, II to IV arteritis level with intermittent limping, under knee femoro popliteal bypass indication.

Available saphenous vein, no major trophic trouble, no contra indication to the use of prosthesis.

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-06; Study Completion 2012-06

PRIMARY OUTCOMES:
Bypass permeability during 5 years after surgery, assessed trough Doppler echography

SECONDARY OUTCOMES:
Mortality and morbidity, primary and secondary permeability, quality of life, leg salvage, cost/benefit ratio.. All patients will be followed up at 1, 3, 6, and 12 months and each year during 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Bordenave, MD-PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Jacques Demotes-Mainard, MD-PhD, Study Chair — CIC INSERM-CHU de Bordeaux
Locations (1):
- Service de chirurgie vasculaire, Hôpital Pellegrin, Place Amélie Raba Léon, Bordeaux, France